CLINICAL TRIAL: NCT07171346
Title: Effects on Patient Outcomes With Post-Operative Use of Zynex Neuromuscular Electrical Stimulation (NMES): Zynex-25
Brief Title: Post Operative Use of Neuromuscular Electrical Stimulation (NMES) Device for ACLR Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Scott Mullen, Associate Professor Orthopedic Surgery & Sports Medicine, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00161884
Record Dates: First submitted 2025-08-22; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: ACL Reconstruction; ACL Surgery; ACL Injury; Electrotherapy; Muscle Atrophy or Weakness
Keywords: Electrotherapy; muscle strength; ACLR
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Muscular Atrophy; Asthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NMES (Experimental): All participants will use the NMES device in addition to standard rehab protocol
  Interventions: Device: Zynex NexWave Electrotherapy Device

INTERVENTIONS:
Device: Zynex NexWave Electrotherapy Device — All participants will use the NMES device in addition to standard rehabilitation

SUMMARY:
This study is being conducted to learn about how neuromuscular electrical stimulation (NMES) in addition to standard of care aids in the recovery of muscle strength in patients undergoing ACLR procedure.

DETAILED DESCRIPTION:
The addition of neuromuscular electrical stimulation (NMES) to standard ACLR rehabilitation has been demonstrated to improve knee extension and flexion compared to standard treatment only. NMES has also shown improved lower limb loading symmetry, walking velocity, stance time, cadence, maximum voluntary isometric contraction, motor unit behavior, muscle quality, and an increase in absolute muscle strength in functional tests compared to standard care of ACLR recovery. In this study we will be comparing bi-lateral presurgical and post surgical muscle strength symmetry in patients that follow the standard ACLR rehabilitation program and patients that use the NMES in addition to standard rehab.

ELIGIBILITY:
Inclusion Criteria:

* ACLR surgical patients at KUMC sports medicine
* 15 to 50 years old
* BMI between 18 - 30 kg/m2
* No limitations impacting physical function within the last 6 months (not including the ACL injury)

Exclusion Criteria:

* Previous lower limb or spine injury involving surgical treatment
* Prior spine surgery
* Lower limb injury (other than ACL) preventing participation in physical activity for over two weeks in the past 6 months
* Non english speaking
* Vulnerable population, prisoner, or ward of the state

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Bilateral Muscle Symmetry Index | pre-operative to 3 months post-op
  Comparing muscle size strength and function between operative and non-operative limbs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melkerson MN. Combination Neuromuscular Electrical Stimulator, Interferential Stimulator, and Transcutaneous Electrical Nerve Stimulator, Model NexWave. In: Services DoHH, editor. Silver Spring, MD: Food and Drug Administration; 2011.
- [Background] Labanca L, Rocchi JE, Giannini S, Faloni ER, Montanari G, Mariani PP, Macaluso A. Early Superimposed NMES Training is Effective to Improve Strength and Function Following ACL Reconstruction with Hamstring Graft regardless of Tendon Regeneration. J Sports Sci Med. 2022 Feb 15;21(1):91-103. doi: 10.52082/jssm.2022.91. eCollection 2022 Mar. PMID 35250338
- [Background] Snyder-Mackler L, Delitto A, Bailey SL, Stralka SW. Strength of the quadriceps femoris muscle and functional recovery after reconstruction of the anterior cruciate ligament. A prospective, randomized clinical trial of electrical stimulation. J Bone Joint Surg Am. 1995 Aug;77(8):1166-73. doi: 10.2106/00004623-199508000-00004. PMID 7642660
- [Background] Conley CEW, Mattacola CG, Jochimsen KN, Dressler EV, Lattermann C, Howard JS. A Comparison of Neuromuscular Electrical Stimulation Parameters for Postoperative Quadriceps Strength in Patients After Knee Surgery: A Systematic Review. Sports Health. 2021 Mar;13(2):116-127. doi: 10.1177/1941738120964817. Epub 2021 Jan 11. PMID 33428557
- [Background] Paternostro-Sluga T, Fialka C, Alacamliogliu Y, Saradeth T, Fialka-Moser V. Neuromuscular electrical stimulation after anterior cruciate ligament surgery. Clin Orthop Relat Res. 1999 Nov;(368):166-75. PMID 10613165
- [Background] Jo HD, Kim MK. Effects of neuromuscular electrical stimulation on neuromuscular function and muscle quality in patient following anterior cruciate ligament reconstruction. J Exerc Rehabil. 2025 Apr 30;21(2):79-91. doi: 10.12965/jer.2550086.043. eCollection 2025 Apr. PMID 40351372
- [Background] Snyder-Mackler L, Ladin Z, Schepsis AA, Young JC. Electrical stimulation of the thigh muscles after reconstruction of the anterior cruciate ligament. Effects of electrically elicited contraction of the quadriceps femoris and hamstring muscles on gait and on strength of the thigh muscles. J Bone Joint Surg Am. 1991 Aug;73(7):1025-36. PMID 1874764
- [Background] Lepley LK, Wojtys EM, Palmieri-Smith RM. Combination of eccentric exercise and neuromuscular electrical stimulation to improve quadriceps function post-ACL reconstruction. Knee. 2015 Jun;22(3):270-7. doi: 10.1016/j.knee.2014.11.013. Epub 2014 Dec 10. PMID 25819154
- [Background] Makihara Y, Nishino A, Fukubayashi T, Kanamori A. Decrease of knee flexion torque in patients with ACL reconstruction: combined analysis of the architecture and function of the knee flexor muscles. Knee Surg Sports Traumatol Arthrosc. 2006 Apr;14(4):310-7. doi: 10.1007/s00167-005-0701-2. Epub 2005 Oct 6. PMID 16208458
- [Background] Konrath JM, Vertullo CJ, Kennedy BA, Bush HS, Barrett RS, Lloyd DG. Morphologic Characteristics and Strength of the Hamstring Muscles Remain Altered at 2 Years After Use of a Hamstring Tendon Graft in Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2016 Oct;44(10):2589-2598. doi: 10.1177/0363546516651441. Epub 2016 Jul 18. PMID 27432052
- [Background] Nomura Y, Kuramochi R, Fukubayashi T. Evaluation of hamstring muscle strength and morphology after anterior cruciate ligament reconstruction. Scand J Med Sci Sports. 2015 Jun;25(3):301-7. doi: 10.1111/sms.12205. Epub 2014 Mar 20. PMID 24646218
- [Background] Currier DP, Ray JM, Nyland J, Rooney JG, Noteboom JT, Kellogg R. Effects of electrical and electromagnetic stimulation after anterior cruciate ligament reconstruction. J Orthop Sports Phys Ther. 1993 Apr;17(4):177-84. doi: 10.2519/jospt.1993.17.4.177. PMID 8467342
- [Background] Heidland A, Fazeli G, Klassen A, Sebekova K, Hennemann H, Bahner U, Di Iorio B. Neuromuscular electrostimulation techniques: historical aspects and current possibilities in treatment of pain and muscle waisting. Clin Nephrol. 2013 Jan;79 Suppl 1:S12-23. PMID 23249528
- See also: Zynex NexWave Device — https://www.zynex.com/products/nexwave/